CLINICAL TRIAL: NCT03199053
Title: A 26 Week, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Parallel Group, Phase 3 Trial With a 26 Week Safety Extension Period Evaluating the Safety and Efficacy of Dapagliflozin 5 and 10 mg, and Saxagliptin 2.5 and 5 mg in Pediatric Patients With Type 2 Diabetes Mellitus Who Are Between 10 and Below 18 Years of Age
Brief Title: Study to Evaluate Safety and Efficacy of Dapagliflozin and Saxagliptin in Patients With Type 2 Diabetes Mellitus (T2DM) Aged 10 to Below 18 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1680C00019; 2015-005042-66 (EudraCT Number)
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; saxagliptin

STUDY DESIGN:
Intervention Model Description: Eligible subjects with HbA1c of 6.5% to 10.5% at screening will be randomized 1:1:1 to receive dapagliflozin 5 mg, saxagliptin 2.5 mg, or placebo. Blinded HbA1c assessment will be performed at Week 12. All subjects with Week 12 HbA1c < 7% will remain on previously assigned randomized treatment. Subjects taking dapagliflozin with Week 12 HbA1c ≥ 7% will be re-randomized in a 1:1 ratio to continue on the low-dose treatment (dapagliflozin 5 mg) or up titrate to the high-dose treatment (dapagliflozin 10 mg). Subjects taking saxagliptin with Week 12 HbA1c ≥ 7% will be re-randomized in a 1:1 ratio to continue on the low-dose treatment (saxagliptin 2.5 mg) or up-titrate to the high-dose treatment (saxagliptin 5 mg). Subjects taking placebo with Week 12 HbA1c ≥ 7% will continue on placebo treatment. All placebo subjects and all subjects taking saxagliptin or dapagliflozin with HbA1c < 7% at Week 12 will go through a dummy 2nd randomization process for maintaining the blinding.
Who Masked: Participant, Investigator
Masking Description: sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Low dose Dapagliflozin (Experimental): Oral route. Start with a low dose of dapagliflozin administered once daily and remain on the low dose regardless of your HbA1c at week 12.
  Interventions: Drug: Dapagliflozin
- Low dose/high dose Dapagliflozin (Experimental): Oral route. Start with a low dose of Dapagliflozin administered once daily and up titrate to the high dose Dapagliflozin administered once daily if HbA1c >= 7% at week 12
  Interventions: Drug: Dapagliflozin
- Low dose Saxagliptin (Experimental): Oral route. Start with a low dose of saxagliptin administered once daily and remain on the low dose regardless of your HbA1c at week 12
  Interventions: Drug: Saxagliptin
- Low dose/high dose Saxagliptin (Experimental): Oral route. Start with a low dose of saxagliptin administered once daily and up titrate to the high dose if HbA1c >= 7% at week 12
  Interventions: Drug: Saxagliptin
- Placebo arm (Placebo Comparator): Oral route. Placebo tablets administered for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 5mg , Once daily Tablets, Oral, 10mg, Once daily
  Other Names: Forxiga
  Arms: Low dose Dapagliflozin; Low dose/high dose Dapagliflozin
Drug: Saxagliptin — Tablets, Oral, 2.5mg Once daily Tablets, Oral, 5mg, Once daily
  Other Names: Onglyza
  Arms: Low dose Saxagliptin; Low dose/high dose Saxagliptin
Drug: Placebo — Matching placebo to dapagliflozin 5mg and 10 mg/saxagliptin 2.5 mg and 5 mg, Tablets, oral, Once daily
  Arms: Placebo arm

SUMMARY:
The primary objective of this study is to determine if there will be a greater mean reduction from baseline in glycated hemoglobin (HbA1c) achieved after 26 weeks of oral double-blind add-on therapy of dapagliflozin or saxagliptin compared to placebo in paediatric T2DM patients with HbA1c levels of 6.5 to 10.5% on diet and exercise and metformin, insulin, or metformin plus insulin.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Target Population
* Previously diagnosed with Type 2 Diabetes Mellitus by World Health Organization/ADA criteria
* HbA1c between 6.5% and 10.5% obtained at screening.
* Currently on diet and exercise and stable dose of at least 1000 mg metformin (IR or XR) for a minimum of 8 weeks, or stable dose of insulin for a minimum of 8 weeks, or a stable combination of at least 1000 mg metformin (IR or XR) and insulin for a minimum of 8 weeks prior to randomization. For those children on insulin, investigators will confirm that attempts at removing insulin from the subject's therapeutic regimen had been previously made but had not been successful.
* Age and Reproductive Status
* Male and female patients eligible if 10 years of age, up to but not including 18 years of age at the time of enrollment/screening. At least 30% of total subjects will be between the ages of 10 and 14 years and at least one third, but no more than two thirds, female subjects.
* Women of childbearing potential must have a negative pregnancy test within 24 hours prior to the start of study drug.
* Women must not be breastfeeding.
* Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drugs: saxagliptin, and dapagliflozin, plus 5 half-lives of study drugs or 30 days (whichever is longer), plus 30 days (duration of ovulatory cycle) for a total of 60 days post treatment completion.

Exclusion Criteria:

* Target Disease Exceptions
* Presence of Type 1 diabetes, as demonstrated by Preexisting diagnosis of Type 1 diabetes,
* Previous diagnosis of monogenic etiology of Type 2 diabetes
* Diabetes ketoacidosis (DKA) within 6 months of screening
* Current use of the following medications for the treatment of diabetes, or use within the specified timeframe prior to screening for the main study:
* Eight weeks: sulfonylureas, alpha glucosidase inhibitors, metiglinide, oral or injectable incretins or incretin mimetics, other antidiabetes medications not otherwise specified.
* Sixteen weeks: thiazolidinediones, DPP-4 inhibitors (with no reported medication related AEs related to DPP-4 inhibitors), sodium glucose cotransporter-2 (SGLT-2) inhibitors (with no reported medication related AEs related to SGLT-2 inhibitors)
* Initiation or discontinuation of prescription or non-prescription weight loss drugs within 8 weeks of screening. Use of prescription or non-prescription weight loss drugs must be stable during the study.
* Medical History and Concurrent Diseases
* Pregnant, positive serum pregnancy test, planning to become pregnant during the clinical trials, or breastfeeding
* History of unstable or rapidly progressive renal disease
* History of unresolved vesico-ureteral reflux
* History of or current, acute or chronic pancreatitis
* History of hemoglobinopathy, with the exception of sickle cell trait or thalassemia minor; or chronic or recurrent hemolysis
* Malignancy within 5 years of the screening visit (with the exception of treated basal cell or treated squamous cell carcinoma)
* Replacement or chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid taken for > 4 weeks within 3 months prior to the Day 1 visit
* Physical and Laboratory Test Findings
* Abnormal renal function,
* An abnormal thyroid-stimulating hormone (TSH) value at enrollment will be further evaluated for free T4. Subjects with abnormal free T4 values will be excluded.
* Hematuria (confirmed by microscopy at screening) with no explanation as judged by the Investigator up to randomization.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2× upper limit of normal (ULN), or clinically significant hepatic disease.
* Serum total bilirubin (TB) > 2x ULN unless exclusively caused by Gilbert's syndrome
* Positive serologic evidence of current infectious liver disease including anti hepatitis A virus (HAV) (IgM), hepatitis B surface antigen (HBsAg), or anti hepatitis C virus (HCV). Patients who have isolated positive anti-hepatitis B surface antibodies may be included.
* Anemia of any etiology
* Volume-depleted subjects.
* Allergies and Adverse Drug Reaction
* Known allergy, sensitivity or contraindication to any study drug or its excipient/vehicle
* Other Exclusion Criteria
* Subject is currently abusing alcohol or other drugs or has done so within the last 6 months prior to the screening visit.
* Prisoners or subjects who are involuntarily incarcerated. (Note: under certain specific circumstances a person who has been imprisoned may be included or permitted to continue as a subject. Strict conditions apply and Sponsor/designee approval is required.)
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
* Psychiatric or cognitive disorder that will, in the opinion of investigators, limit the subject's ability to comply with the study medications and monitoring.
* Subjects who have contraindications to therapy as outlined in the saxagliptin and dapagliflozin Investigator Brochure or local package inserts.
* Participation and receiving IP in another clinical study during the prior 3 months

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 256 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (107):
- United States (15):
  - Research Site, Sacramento, California
  - Research Site, New Haven, Connecticut
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Neptune City, New Jersey
  - Research Site, Memphis, Tennessee
  - Research Site, Edinburg, Texas
  - Research Site, Harlingen, Texas
  - Research Site, McAllen, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, San Miguel de Tucumán
- Research Site, Blacktown, Australia
- Brazil (8):
  - Research Site, Brasília
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Santa Maria
  - Research Site, São Paulo
- Research Site, Montreal, Quebec, Canada
- Research Site, Santiago, Chile
- Colombia (2):
  - Research Site, Armenia
  - Research Site, Barranquilla
- Research Site, Tampere, Finland
- India (12):
  - Research Site, Ahmedabad
  - Research Site, Aurangabad
  - Research Site, Bangalore
  - Research Site, Bikaner
  - Research Site, Chandigarh
  - Research Site, Coimbatore
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Kozhikode
  - Research Site, Nashik
  - Research Site, Pune
  - Research Site, Visakhapatnam
- Research Site, Haifa, Israel
- Italy (3):
  - Research Site, Ancona
  - Research Site, Napoli
  - Research Site, Roma
- Malaysia (12):
  - Research Site, George Town
  - Research Site, Ipoh
  - Research Site, Johor Bahru
  - Research Site, Klang
  - Research Site, Kota Kinabalu
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Malacca
  - Research Site, Putrajaya
  - Research Site, Seremban
  - Research Site, Seri Manjung
  - Research Site, Taiping
- Mexico (15):
  - Research Site, Boca del Rio
  - Research Site, Celaya
  - Research Site, Ciudad Madero
  - Research Site, Cuernavaca
  - Research Site, Culiacán
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Juriquilla
  - Research Site, Mérida
  - Research Site, México
  - Research Site, México, D.F.
  - Research Site, Monterrey
  - Research Site, San Juan del Río
  - Research Site, Veracruz
  - Research Site, Zapopan
- New Zealand (3):
  - Research Site, Grafton
  - Research Site, Tauranga
  - Research Site, Wellington
- Philippines (2):
  - Research Site, Quezon City
  - Research Site, San Fernando City
- Research Site, Warsaw, Poland
- Russia (3):
  - Research Site, Izhevsk
  - Research Site, Moscow
  - Research Site, Ufa
- South Korea (3):
  - Research Site, Daejeon
  - Research Site, Incheon
  - Research Site, Wŏnju
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Hat Yai
- Turkey (Türkiye) (8):
  - Research Site, Aydin
  - Research Site, Bursa
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Kurupelit
  - Research Site, Manisa
- Ukraine (3):
  - Research Site, Dnipro
  - Research Site, Kyiv
  - Research Site, Vinnytsia
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, London
  - Research Site, Middlesbrough
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Shehadeh N, Barrett T, Galassetti P, Karlsson C, Monyak J, Iqbal N, Tamborlane WV. Dapagliflozin or Saxagliptin in Pediatric Type 2 Diabetes. NEJM Evid. 2023 Dec;2(12):EVIDoa2300210. doi: 10.1056/EVIDoa2300210. Epub 2023 Oct 4. PMID 38320500
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1680C00019&attachmentIdentifier=9f610176-081e-4659-a955-31192c46471e&fileName=CSR_Synopsis_Redacted_pdfa.pdf&versionIdentifier=
- See also: SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1680C00019&attachmentIdentifier=a8045694-354d-4408-bff7-6fee81e69119&fileName=SAP_Redacted_pdfa.pdf&versionIdentifier=
- See also: CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1680C00019&attachmentIdentifier=ffb4f464-404c-4c9e-8a5d-1366c1c38e5a&fileName=CSP_Redacted_pdfa.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 245 patients were randomised from 94 sites in 21 countries. Participants were initially randomised in a 1:1:1 ratio to receive dapagliflozin 5 mg, saxagliptin 2.5 mg, or placebo.
Pre-assignment Details: An initial 26-week short-term (ST) period was followed by a 26-week long-term (LT) safety extension period. The study drug was discontinued at Week 52, after which participants continued in the Non-treatment Follow-up Period until Week 104.
  Of the 256 participants enrolled, 11 were excluded from analysis due to GCP considerations at the site they originated from (see limitations and caveats for further details).
Groups:
- Dapagliflozin: Participants were randomised to receive dapagliflozin 5 mg administered orally once daily (low-dose). At Week 14, participants with Week 12 glycated haemoglobin (HbA1c) values < 7% remained on low-dose dapagliflozin. Participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to dapagliflozin 10 mg administered orally once daily (high-dose).
  After completion of the ST treatment period, participants could enter the LT treatment period. Participants who were receiving background medication with insulin only or insulin and metformin (not eligible for the third randomisation) continued with their randomised study drug assigned after the second randomisation.
  A subset of eligible participants (on background treatment with metformin only and who had HbA1c < 7.5% at Week 26 or Week 32) were grouped into 2 separate strata for saxagliptin and dapagliflozin, and then randomised 1:1 within each of the strata to either continue or discontinue background medication with metformin at either Week 32 or Week 40. For participants randomised to withdraw background treatment with metformin, those receiving high-dose treatment continued to receive high-dose treatment, whereas those currently receiving low-dose treatment had their doses uptitrated to high-dose treatment. Participants who were randomized to continue background medication with metformin continued with their current dose of dapagliflozin.
- Saxagliptin: Participants were randomised to receive saxagliptin 2.5 mg administered orally once daily (low-dose). At Week 14, participants with Week 12 HbA1c values < 7% remained on low-dose saxagliptin. Participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to saxagliptin 5 mg administered orally once daily (high-dose).
  After completion of the ST treatment period, participants could enter the LT treatment period. Participants who were receiving background medication with insulin only or insulin and metformin (not eligible for the third randomisation) continued with their randomised study drug assigned after the second randomisation.
  A subset of eligible participants (on background treatment with metformin only and who had HbA1c < 7.5% at Week 26 or Week 32) were grouped into 2 separate strata for saxagliptin and dapagliflozin, and then randomised 1:1 within each of the strata to either continue or discontinue background medication with metformin at either Week 32 or Week 40. For participants randomised to withdraw background treatment with metformin, those receiving high-dose treatment continued to receive high-dose treatment, whereas those currently receiving low-dose treatment had their doses uptitrated to high-dose treatment. Participants who were randomized to continue background medication with metformin continued with their current dose of saxagliptin.
- Placebo: Participants were randomised to receive placebo administered orally once daily. At Week 14, all participants continued on placebo. To maintain blinding, all participants underwent a dummy second randomisation process that was undistinguishable from the actual second randomisation.
  After completion of the ST treatment period, participants could enter the LT treatment period. Participants who were receiving background medication with insulin only or insulin and metformin (not eligible for the third randomisation) continued with their randomised study drug assigned after the second randomisation.
  At either Week 32 or Week 40 eligible participants receiving placebo (on background treatment with metformin only and who had HbA1c < 7.5% at Week 26 or Week 32) were randomised 1:1:1 to either withdraw background medication with metformin and switch to active treatment with either saxagliptin 5 mg or dapagliflozin 10 mg or to remain on background medication with metformin and continue with placebo.
Period: ST Period
Arm/Group | Dapagliflozin | Saxagliptin | Placebo
Started | 81 | 88 | 76
Week 14 no Uptitration Randomisation (Excluded from Uptitration Randomised Participants Data Set.) | 39 | 36 | 0
Week 14 Uptitration Randomisation (Included in Uptitration Randomised Participants Data Set.) | 42 | 52 | 0
Completed | 76 | 83 | 68
Not Completed | 5 | 5 | 8
Not completed — Withdrawal by Subject | 2 | 4 | 6
Not completed — Withdrawal by parent/guardian | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1
Period: LT Period
Arm/Group | Dapagliflozin | Saxagliptin | Placebo
Started | 76 | 83 | 68
Randomised Withdrawal Patients Data Set | 13 | 25 | 8
Excluded From Randomised Withdrawal Patients Data Set | 68 | 63 | 68
Randomised to Continue Metformin (Pre-specified in the statistical analysis plan, only participants who continued or discontinued metformin after the third randomization were collected.) | 6 | 12 | 2
Randomised Metformin Withdrawal (Pre-specified in the statistical analysis plan, only participants who continued or discontinued metformin after the third randomization were collected.) | 7 | 13 | 6
Completed | 75 | 79 | 61
Not Completed | 1 | 4 | 7
Not completed — Withdrawal by Subject | 1 | 3 | 3
Not completed — Withdrawal by parent/guardian | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Miscellaneous | 0 | 0 | 2
Period: Non-treatment Follow-up Period
Arm/Group | Dapagliflozin | Saxagliptin | Placebo
Started | 74 (One participant withdrew following the LT Period, prior to starting the Non-treatment Follow-up Period.) | 77 (Two participants withdrew following the LT Period, prior to starting the Non-treatment Follow-up Period.) | 59 (Two participants withdrew following the LT Period, prior to starting the Non-treatment Follow-up Period.)
Completed | 67 | 68 | 52
Not Completed | 7 | 9 | 7
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Withdrawal by parent/guardian | 2 | 3 | 2
Not completed — Lost to Follow-up | 3 | 4 | 5
Not completed — Miscellaneous | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomised Participants Data Set: consisted of all randomised participants who receive at least one dose of study medication during the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Saxagliptin | Placebo | Total
Number analyzed (Participants) | 81 | 88 | 76 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (2.00) | 14.5 (1.75) | 14.7 (1.64) | 14.5 (1.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 53 | 44 | 146
  Male | 32 | 35 | 32 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 43 | 34 | 122
  Not Hispanic or Latino | 36 | 45 | 42 | 123
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 50 | 32 | 124
  Black or African American | 7 | 4 | 3 | 14
  Asian | 18 | 23 | 24 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 3 | 3
  American Indian or Alaska Native | 11 | 7 | 12 | 30
  Other | 3 | 4 | 2 | 9
Mean Baseline HbA1c [Mean (Standard Deviation); unit: Percentage HbA1c] | 8.22 (1.459) | 8.02 (1.431) | 7.96 (1.629) | 8.07 (1.502)

OUTCOME MEASURES:

1. Primary Outcome: Dapagliflozin Versus Placebo: Adjusted Mean Change From Baseline in HbA1c at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline HbA1c as covariate. Missing Week 26 data was handled based on multiple imputation washout (MI-WO) within each arm using the data from placebo participants with Week 26 data.
Time Frame: Baseline and Week 26
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Percentage HbA1c
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 75 | 70
Percentage HbA1c | -0.62 (0.218) | 0.41 (0.218)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Adjusted mean difference = -1.03, 95% CI 2-sided [-1.57 to -0.49], Standard Error of Mean 0.274

2. Primary Outcome: Saxagliptin Versus Placebo: Adjusted Mean Change From Baseline in HbA1c at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline HbA1c as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
Time Frame: Baseline and Week 26
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Percentage HbA1c
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 82 | 70
Percentage HbA1c | 0.06 (0.198) | 0.50 (0.202)
Statistical Analysis 1: Comparison: Saxagliptin vs Placebo; Test type: Superiority; p = 0.078, ANCOVA; Adjusted mean difference = -0.44, 95% CI 2-sided [-0.93 to 0.05], Standard Error of Mean 0.251

3. Secondary Outcome: Dapagliflozin Low-dose/High-dose Versus Placebo (Weighted): Adjusted Mean Change From Baseline in HbA1c at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline HbA1c as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Dapagliflozin participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 0; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 2; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: Randomised Participants Data Set: consisted of all randomised participants who receive at least one dose of study medication during the treatment period. Includes participants with available data only. Data is pooled for Dapagliflozin 5 mg/10 mg and weighted as pre-specified in the statistical analysis plan.
Measure: Mean (Standard Error); unit: Percentage HbA1c
Groups:
- Dapagliflozin 5 mg/10 mg (Weighted): Participants were randomised to receive dapagliflozin 5 mg administered orally once daily (low-dose). At Week 14, participants with Week 12 HbA1c values < 7% remained on low-dose dapagliflozin (weight = 1). Participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment (weight = 0) or to uptitrate to dapagliflozin 10 mg administered orally once daily (high-dose) (weight = 2).
  After completion of the ST treatment period, participants could enter the LT treatment period.
- Placebo (Weight = 1): Participants were randomised to receive placebo administered orally once daily. At Week 14, all participants continued on placebo. To maintain blinding, all participants underwent a dummy second randomisation process that was undistinguishable from the actual second randomisation.
  After completion of the ST treatment period, participants could enter the LT treatment period.
Arm/Group | Dapagliflozin 5 mg/10 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 54 | 70
Percentage HbA1c | -0.42 (0.214) | 0.43 (0.207)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg/10 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.004, ANCOVA; Adjusted mean difference = -0.86, 95% CI 2-sided [-1.44 to -0.27], Standard Error of Mean 0.300

4. Secondary Outcome: Saxagliptin Low-dose/High-dose Versus Placebo (Weighted): Adjusted Mean Change From Baseline in HbA1c at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline HbA1c as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Saxagliptin participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 0; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 2; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: Randomised Participants Data Set: consisted of all randomised participants who receive at least one dose of study medication during the treatment period. Includes participants with available data only. Data is pooled for Saxagliptin 2.5 mg/5 mg and weighted as pre-specified in the statistical analysis plan.
Measure: Mean (Standard Error); unit: Percentage HbA1c
Groups:
- Saxagliptin 2.5 mg/5 mg (Weighted): Participants were randomised to receive saxagliptin 2.5 mg administered orally once daily (low-dose). At Week 14, participants with Week 12 HbA1c values < 7% remained on low-dose saxagliptin (weight = 1). Participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment (weight = 0) or to uptitrate to saxagliptin 5 mg administered orally once daily (high-dose) (weight = 2).
  After completion of the ST treatment period, participants could enter the LT treatment period.
Arm/Group | Saxagliptin 2.5 mg/5 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 58 | 70
Percentage HbA1c | -0.04 (0.190) | 0.47 (0.200)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg/5 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.067, ANCOVA; Adjusted mean difference = -0.51, 95% CI 2-sided [-1.05 to 0.04], Standard Error of Mean 0.277

5. Secondary Outcome: Dapagliflozin Low-dose Versus Placebo (Weighted): Adjusted Mean Change From Baseline in HbA1c at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline HbA1c as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Dapagliflozin participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 2; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 0; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Percentage HbA1c
Arm/Group | Dapagliflozin 5 mg/10 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 56 | 70
Percentage HbA1c | -0.79 (0.202) | 0.40 (0.205)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg/10 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p < 0.001, ANCOVA; Adjusted mean difference = -1.19, 95% CI 2-sided [-1.76 to -0.62], Standard Error of Mean 0.290

6. Secondary Outcome: Saxagliptin Low-dose Versus Placebo (Weighted): Adjusted Mean Change From Baseline in HbA1c at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline HbA1c as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Saxagliptin participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 2; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 0; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Percentage HbA1c
Arm/Group | Saxagliptin 2.5 mg/5 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 57 | 70
Percentage HbA1c | 0.07 (0.188) | 0.47 (0.194)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg/5 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.146, ANCOVA; Adjusted mean difference = -0.39, 95% CI 2-sided [-0.92 to 0.14], Standard Error of Mean 0.270

7. Secondary Outcome: Dapagliflozin Versus Placebo: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline FPG as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
Time Frame: Baseline and Week 26
Population: Randomised Participants Data Set: consisted of all randomised participants who receive at least one dose of study medication during the treatment period. Includes participants with available data only.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 75 | 68
mmol/L | -0.57 (0.374) | 0.51 (0.384)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority; p = 0.024, ANCOVA; Adjusted mean difference = -1.08, 95% CI 2-sided [-2.02 to -0.14], Standard Error of Mean 0.479

8. Secondary Outcome: Saxagliptin Versus Placebo: Adjusted Mean Change From Baseline in FPG at Week 26
Description: as for outcome 7
Time Frame: Baseline and Week 26
Population: as for outcome 7
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 80 | 68
mmol/L | 0.08 (0.413) | 0.19 (0.428)
Statistical Analysis 1: Comparison: Saxagliptin vs Placebo; Test type: Superiority; p = 0.833, ANCOVA; Adjusted mean difference = -0.11, 95% CI 2-sided [-1.15 to 0.92], Standard Error of Mean 0.528

9. Secondary Outcome: Dapagliflozin Low-dose/High-dose Versus Placebo (Weighted): Adjusted Mean Change From Baseline in FPG at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline FPG as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Dapagliflozin participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 0; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 2; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Dapagliflozin 5 mg/10 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 54 | 68
mmol/L | -0.34 (0.365) | 0.70 (0.369)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg/10 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.047, ANCOVA; Adjusted mean difference = -1.04, 95% CI 2-sided [-2.07 to -0.01], Standard Error of Mean 0.525

10. Secondary Outcome: Saxagliptin Low-dose/High-dose Versus Placebo (Weighted): Adjusted Mean Change From Baseline in FPG at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline FPG as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Saxagliptin participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 0; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 2; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin 2.5 mg/5 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 57 | 68
mmol/L | 0.18 (0.331) | 0.73 (0.359)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg/5 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.268, ANCOVA; Adjusted mean difference = -0.54, 95% CI 2-sided [-1.50 to 0.42], Standard Error of Mean 0.490

11. Secondary Outcome: Dapagliflozin Low-dose Versus Placebo (Weighted): Adjusted Mean Change From Baseline in FPG at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline FPG as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Dapagliflozin participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 2; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 0; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Dapagliflozin 5 mg/10 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 56 | 68
mmol/L | -0.56 (0.347) | 0.56 (0.363)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg/10 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.026, ANCOVA; Adjusted mean difference = -1.12, 95% CI 2-sided [-2.11 to -0.13], Standard Error of Mean 0.505

12. Secondary Outcome: Saxagliptin Low-dose Versus Placebo (Weighted): Adjusted Mean Change From Baseline in FPG at Week 26
Description: Data was analysed with an ANCOVA model with treatment, sex, age group and background antidiabetes medication as factors and Baseline FPG as covariate. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Saxagliptin participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 2; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 0; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin 2.5 mg/5 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 55 | 68
mmol/L | 0.63 (0.424) | 0.34 (0.446)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg/5 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.644, ANCOVA; Adjusted mean difference = 0.29, 95% CI 2-sided [-0.92 to 1.50], Standard Error of Mean 0.618

13. Secondary Outcome: Percentage of Participants With Baseline HbA1c ≥ 7% Who Achieved HbA1c < 7% at Week 26
Description: A logistic regression model adjusting for sex, age group, background antidiabetes medication and Baseline HbA1c was used. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
Time Frame: Baseline and Week 26
Population: Randomised Participants Data Set: consisted of all randomised participants who receive at least one dose of study medication during the treatment period. Includes participants with Baseline HbA1c >= 7% and available data only.
Measure: Number; unit: Percentage of participants
Arm/Group | Dapagliflozin | Saxagliptin | Placebo
Number analyzed (Participants) | 64 | 61 | 50
Percentage of participants | 26.6 | 21.3 | 10.0
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority; p = 0.019, Regression, Logistic; Adjusted Odds Ratio = 3.8, 95% CI 2-sided [1.2 to 11.7]
Statistical Analysis 2: Comparison: Saxagliptin vs Placebo; Test type: Superiority; p = 0.114, Regression, Logistic; Adjusted Odds Ratio = 2.6, 95% CI 2-sided [0.8 to 8.6]

14. Secondary Outcome: Low-dose/High-dose Versus Placebo (Weighted): Percentage of Participants With Baseline HbA1c ≥ 7% Who Achieved HbA1c < 7% at Week 26
Description: A weighted logistic regression model adjusting for sex, age group, background antidiabetes medication and Baseline HbA1c was used. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 0; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 2; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: Randomised Participants Data Set: consisted of all randomised participants who receive at least one dose of study medication during the treatment period. Includes participants with Baseline HbA1c >= 7% and available data only. Data is pooled for Dapagliflozin 5 mg/10 mg and Saxagliptin 2.5 mg/5 mg and weighted as pre-specified in the statistical analysis plan.
Measure: Number; unit: Percentage of participants
Arm/Group | Dapagliflozin 5 mg/10 mg (Weighted) | Saxagliptin 2.5 mg/5 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 44 | 41 | 50
Percentage of participants | 27.3 | 24.4 | 10.0
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg/10 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.042, Weighted Logistic Regression; Adjusted Odds Ratio = 3.5, 95% CI 2-sided [1.0 to 11.4]
Statistical Analysis 2: Comparison: Saxagliptin 2.5 mg/5 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.175, Weighted Logistic Regression; Adjusted Odds Ratio = 2.3, 95% CI 2-sided [0.7 to 7.4]

15. Secondary Outcome: Low-dose Versus Placebo (Weighted): Percentage of Participants With Baseline HbA1c ≥ 7% Who Achieved HbA1c < 7% at Week 26
Description: A weighted logistic regression model adjusting for sex, age group, background antidiabetes medication and Baseline HbA1c was used. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
  Participants were weighted as follows: participants who had HbA1c < 7% at Week 12 and remained on low-dose were assigned a weight of 1; participants who had HbA1c >= 7% at Week 12 and continued on the low-dose were assigned a weight of 2; participants who had HbA1c >= 7% at Week 12 and received the high-dose were assigned a weight of 0; all participants who do not undergo second randomisation were assigned a weight of 1. Placebo participants were assigned a weight of 1.
Time Frame: Baseline and Week 26
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Dapagliflozin 5 mg/10 mg (Weighted) | Saxagliptin 2.5 mg/5 mg (Weighted) | Placebo (Weight = 1)
Number analyzed (Participants) | 45 | 38 | 50
Percentage of participants | 35.6 | 28.9 | 10.0
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg/10 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.009, Weighted Logistic Regression; Adjusted Odds Ratio = 4.4, 95% CI 2-sided [1.4 to 13.2]
Statistical Analysis 2: Comparison: Saxagliptin 2.5 mg/5 mg (Weighted) vs Placebo (Weight = 1); Test type: Superiority; p = 0.042, Weighted Logistic Regression; Adjusted Odds Ratio = 3.8, 95% CI 2-sided [1.1 to 13.5]

16. Secondary Outcome: Low-dose Versus Uptitration to the High Dose: Adjusted Mean Change From Baseline in HbA1c at Week 26
Description: as for outcome 2
Time Frame: Baseline and Week 26
Population: Uptitration Randomised Participants Data Set: consisted of the subset of randomised participants who were up-titration randomised because their HbA1c is greater than or equal to 7% at Week 12 (regardless of rescue medication initiation). Includes participants with available data only.
Measure: Mean (Standard Error); unit: Percentage HbA1c
Groups:
- Dapagliflozin 10 mg: Participants were randomised to receive dapagliflozin 5 mg administered orally once daily (low-dose). At Week 14, participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to dapagliflozin 10 mg administered orally once daily (high-dose).
  After completion of the ST treatment period, participants could enter the LT treatment period.
- Dapagliflozin 5 mg: Participants were randomised to receive dapagliflozin 5 mg administered orally once daily (low-dose). At Week 14, participants with Week 12 HbA1c values < 7% remained on low-dose dapagliflozin. Participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to dapagliflozin 10 mg administered orally once daily (high-dose).
  After completion of the ST treatment period, participants could enter the LT treatment period.
- Saxagliptin 5 mg: Participants were randomised to receive saxagliptin 2.5 mg administered orally once daily (low-dose). At Week 14, participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to saxagliptin 5 mg administered orally once daily (high-dose).
  After completion of the ST treatment period, participants could enter the LT treatment period.
- Saxagliptin 2.5 mg: Participants were randomised to receive saxagliptin 2.5 mg administered orally once daily (low-dose). At Week 14, participants with Week 12 HbA1c values < 7% remained on low-dose saxagliptin. Participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to saxagliptin 5 mg administered orally once daily (high-dose).
  After completion of the ST treatment period, participants could enter the LT treatment period.
Arm/Group | Dapagliflozin 10 mg | Dapagliflozin 5 mg | Saxagliptin 5 mg | Saxagliptin 2.5 mg
Number analyzed (Participants) | 19 | 21 | 25 | 24
Percentage HbA1c | -0.74 (0.368) | -0.71 (0.384) | -0.16 (0.361) | 0.07 (0.372)
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Dapagliflozin 5 mg; Test type: Superiority; p = 0.955, ANCOVA; Adjusted mean difference = -0.03, 95% CI 2-sided [-1.00 to 0.94], Standard Error of Mean 0.496
Statistical Analysis 2: Comparison: Saxagliptin 5 mg vs Saxagliptin 2.5 mg; Test type: Superiority; p = 0.640, ANCOVA; Adjusted mean difference = -0.23, 95% CI 2-sided [-1.20 to 0.74], Standard Error of Mean 0.495

17. Secondary Outcome: Low-dose Versus Uptitration to the High Dose: Adjusted Mean Change From Baseline in FPG at Week 26
Description: as for outcome 7
Time Frame: Baseline and Week 26
Population: as for outcome 16
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Dapagliflozin 10 mg | Dapagliflozin 5 mg | Saxagliptin 5 mg | Saxagliptin 2.5 mg
Number analyzed (Participants) | 19 | 21 | 25 | 23
mmol/L | -1.62 (0.689) | -0.98 (0.683) | -2.38 (0.734) | -0.56 (0.763)
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Dapagliflozin 5 mg; Test type: Superiority; p = 0.476, ANCOVA; Adjusted mean difference = -0.64, 95% CI 2-sided [-2.39 to 1.12], Standard Error of Mean 0.896
Statistical Analysis 2: Comparison: Saxagliptin 5 mg vs Saxagliptin 2.5 mg; Test type: Superiority; p = 0.075, ANCOVA; Adjusted mean difference = -1.81, 95% CI 2-sided [-3.81 to 0.18], Standard Error of Mean 1.017

18. Secondary Outcome: Dapagliflozin Low-dose Versus Uptitration to the High Dose: Percentage of Participants With Baseline HbA1c ≥ 7% Who Achieved HbA1c < 7% at Week 26
Description: A Fisher's exact test was used and unadjusted difference in percentage of participants and Clopper-Pearson CIs presented using imputed data. Missing Week 26 data was handled based on MI-WO within each arm using the data from placebo participants with Week 26 data.
Time Frame: Baseline and Week 26
Population: as for outcome 16
Measure: Number; unit: Percentage of participants
Arm/Group | Dapagliflozin 10 mg | Dapagliflozin 5 mg
Number analyzed (Participants) | 19 | 20
Percentage of participants | 5.3 | 25.0
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Dapagliflozin 5 mg; Test type: Superiority; p = 0.182, Fisher Exact; Unadjusted Difference in Percentage = -19.7, 95% CI 2-sided [-44.5 to 5.7]

19. Secondary Outcome: Saxagliptin Low-dose Versus Uptitration to the High Dose: Percentage of Participants With Baseline HbA1c ≥ 7% Who Achieved HbA1c < 7% at Week 26
Description: as for outcome 18
Time Frame: Baseline and Week 26
Population: as for outcome 16
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 5 mg | Saxagliptin 2.5 mg
Number analyzed (Participants) | 23 | 20
Percentage of participants | 8.7 | 15.0
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Saxagliptin 2.5 mg; Test type: Superiority; p = 0.650, Fisher Exact; Unadjusted Difference in Percentage = -6.3, 95% CI 2-sided [-29.8 to 16.5]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to Week 104 Serious and other AEs: Up to 52 Weeks + 30 days (Week 56)
Description: Treated Participants Data Set: consisted of all participants who received at least one dose of study medication. As pre-specified in the statistical analysis plan, adverse events data for participants continuing on metformin following third randomization and for participants who were not eligible for the third randomization were not collected separately.
Groups:
- Weeks 1 to 14: Dapagliflozin 5 mg: Participants were randomised to receive dapagliflozin 5 mg administered orally once daily (low-dose).
- Weeks 14 to 26: Dapagliflozin 5 mg: At Week 14, participants with Week 12 HbA1c values < 7% remained on low-dose dapagliflozin. Participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to dapagliflozin 10 mg administered orally once daily (high-dose).
- Weeks 14 to 26: Dapagliflozin 10 mg: At Week 14, participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to dapagliflozin 10 mg administered orally once daily (high-dose).
- Weeks 26 to 56: Dapagliflozin 5 mg; Weeks 26 to 56: Dapagliflozin 10 mg: After completion of the ST treatment period, participants could enter the LT treatment period. Participants who were receiving background medication with insulin only or insulin and metformin (not eligible for the third randomisation) continued with their randomised study drug assigned after the second randomisation.
  A subset of eligible participants (on background treatment with metformin only and who had HbA1c < 7.5% at Week 26 or Week 32) were grouped into 2 separate strata for saxagliptin and dapagliflozin, and then randomised 1:1 within each of the strata to either continue or discontinue background medication with metformin at either Week 32 or Week 40. Participants who were randomized to continue background medication with metformin continued with their current dose of dapagliflozin.
- Weeks 32 or 40 to 56: Dapagliflozin 10 mg + Metformin Withdrawal: After completion of the ST treatment period, participants could enter the LT treatment period.
  A subset of eligible participants (on background treatment with metformin only and who had HbA1c < 7.5% at Week 26 or Week 32) were grouped into 2 separate strata for dapagliflozin, and then randomised 1:1 within each of the strata to either continue or discontinue background medication with metformin at either Week 32 or Week 40. For participants randomised to withdraw background treatment with metformin, those receiving high-dose treatment continued to receive high-dose treatment, whereas those currently receiving low-dose treatment had their doses uptitrated to high-dose treatment.
- Weeks 1 to 14: Saxagliptin 2.5 mg: Participants were randomised to receive saxagliptin 2.5 mg administered orally once daily (low-dose).
- Weeks 14 to 26: Saxagliptin 2.5 mg: At Week 14, participants with Week 12 HbA1c values < 7% remained on low-dose saxagliptin. Participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to saxagliptin 5 mg administered orally once daily (high-dose).
- Weeks 14 to 26: Saxagliptin 5 mg: At Week 14, participants with Week 12 HbA1c values ≥ 7% were re-randomised in a 1:1 ratio to continue on low-dose treatment or to uptitrate to saxagliptin 5 mg administered orally once daily (high-dose).
- Weeks 26 to 56: Saxagliptin 2.5 mg; Weeks 26 to 56: Saxagliptin 5 mg: After completion of the ST treatment period, participants could enter the LT treatment period. Participants who were receiving background medication with insulin only or insulin and metformin (not eligible for the third randomisation) continued with their randomised study drug assigned after the second randomisation.
  A subset of eligible participants (on background treatment with metformin only and who had HbA1c < 7.5% at Week 26 or Week 32) were grouped into 2 separate strata for saxagliptin and dapagliflozin, and then randomised 1:1 within each of the strata to either continue or discontinue background medication with metformin at either Week 32 or Week 40. Participants who were randomized to continue background medication with metformin continued with their current dose of saxagliptin.
- Weeks 32 or 40 to 56: Saxagliptin 5 mg + Metformin Withdrawal: After completion of the ST treatment period, participants could enter the LT treatment period.
  A subset of eligible participants (on background treatment with metformin only and who had HbA1c < 7.5% at Week 26 or Week 32) were grouped into 2 separate strata for saxagliptin, and then randomised 1:1 within each of the strata to either continue or discontinue background medication with metformin at either Week 32 or Week 40. For participants randomised to withdraw background treatment with metformin, those receiving high-dose treatment continued to receive high-dose treatment, whereas those currently receiving low-dose treatment had their doses uptitrated to high-dose treatment.
- Weeks 1 to 14: Placebo: Participants were randomised to receive placebo administered orally once daily.
- Weeks 14 to 26: Placebo: At Week 14, all participants continued on placebo. To maintain blinding, all participants underwent a dummy second randomisation process that was undistinguishable from the actual second randomisation.
- Weeks 26 to 32 or 40: Placebo: After completion of the ST treatment period, participants could enter the LT treatment period.
  Participants who were receiving background medication with insulin only or insulin and metformin (not eligible for the third randomisation) continued with their randomised study drug assigned after the second randomisation.
  At either Week 32 or Week 40 eligible participants receiving placebo were randomised 1:1:1 to either withdraw background medication with metformin and switch to active treatment with either saxagliptin 5 mg or dapagliflozin 10 mg or to remain on background medication with metformin and continue with placebo.
- Weeks 32 or 40 to 56: Placebo: Participants who were receiving background medication with insulin only or insulin and metformin (not eligible for the third randomisation) continued with their randomised study drug assigned after the second randomisation.
  At either Week 32 or Week 40 eligible participants receiving placebo were randomised 1:1:1 to either withdraw background medication with metformin and switch to active treatment with either saxagliptin 5 mg or dapagliflozin 10 mg or to remain on background medication with metformin and continue with placebo.
- Weeks 32 or 40 to 56: Placebo to Dapagliflozin 10 mg + Metformin Withdrawal; Weeks 32 or 40 to 56: Placebo to Saxagliptin 5 mg + Metformin Withdrawal: At either Week 32 or Week 40 eligible participants receiving placebo were randomised 1:1:1 to either withdraw background medication with metformin and switch to active treatment with either saxagliptin 5 mg or dapagliflozin 10 mg or to remain on background medication with metformin and continue with placebo.
- Week 56 to 104: Non-treatment Follow-up Period: Safety monitoring continued in the Non-treatment Follow-up Period quarterly between the Week 56 and Week 104 visits.
Arm/Group | Weeks 1 to 14: Dapagliflozin 5 mg | Weeks 14 to 26: Dapagliflozin 5 mg | Weeks 14 to 26: Dapagliflozin 10 mg | Weeks 26 to 56: Dapagliflozin 5 mg | Weeks 26 to 56: Dapagliflozin 10 mg | Weeks 32 or 40 to 56: Dapagliflozin 10 mg + Metformin Withdrawal | Weeks 1 to 14: Saxagliptin 2.5 mg | Weeks 14 to 26: Saxagliptin 2.5 mg | Weeks 14 to 26: Saxagliptin 5 mg | Weeks 26 to 56: Saxagliptin 2.5 mg | Weeks 26 to 56: Saxagliptin 5 mg | Weeks 32 or 40 to 56: Saxagliptin 5 mg + Metformin Withdrawal | Weeks 1 to 14: Placebo | Weeks 14 to 26: Placebo | Weeks 26 to 32 or 40: Placebo | Weeks 32 or 40 to 56: Placebo | Weeks 32 or 40 to 56: Placebo to Dapagliflozin 10 mg + Metformin Withdrawal | Weeks 32 or 40 to 56: Placebo to Saxagliptin 5 mg + Metformin Withdrawal | Week 56 to 104: Non-treatment Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/55 | 0/21 | 0/55 | 0/21 | 0/7 | 0/88 | 0/61 | 0/26 | 0/61 | 0/26 | 0/13 | 0/76 | 0/70 | 0/70 | 0/53 | 0/3 | 0/3 | 0/210
Serious Adverse Events (participants affected / at risk) | 1/81 | 0/55 | 0/21 | 5/55 | 1/21 | 0/7 | 2/88 | 1/61 | 0/26 | 3/61 | 1/26 | 0/13 | 1/76 | 1/70 | 3/70 | 0/53 | 0/3 | 0/3 | 0/210
Other Adverse Events (participants affected / at risk) | 35/81 | 14/55 | 4/21 | 26/55 | 8/21 | 2/7 | 37/88 | 18/61 | 10/26 | 23/61 | 12/26 | 3/13 | 39/76 | 24/70 | 29/70 | 2/53 | 1/3 | 1/3 | 0/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weeks 1 to 14: Dapagliflozin 5 mg (N=81) | Weeks 14 to 26: Dapagliflozin 5 mg (N=55) | Weeks 14 to 26: Dapagliflozin 10 mg (N=21) | Weeks 26 to 56: Dapagliflozin 5 mg (N=55) | Weeks 26 to 56: Dapagliflozin 10 mg (N=21) | Weeks 32 or 40 to 56: Dapagliflozin 10 mg + Metformin Withdrawal (N=7) | Weeks 1 to 14: Saxagliptin 2.5 mg (N=88) | Weeks 14 to 26: Saxagliptin 2.5 mg (N=61) | Weeks 14 to 26: Saxagliptin 5 mg (N=26) | Weeks 26 to 56: Saxagliptin 2.5 mg (N=61) | Weeks 26 to 56: Saxagliptin 5 mg (N=26) | Weeks 32 or 40 to 56: Saxagliptin 5 mg + Metformin Withdrawal (N=13) | Weeks 1 to 14: Placebo (N=76) | Weeks 14 to 26: Placebo (N=70) | Weeks 26 to 32 or 40: Placebo (N=70) | Weeks 32 or 40 to 56: Placebo (N=53) | Weeks 32 or 40 to 56: Placebo to Dapagliflozin 10 mg + Metformin Withdrawal (N=3) | Weeks 32 or 40 to 56: Placebo to Saxagliptin 5 mg + Metformin Withdrawal (N=3) | Week 56 to 104: Non-treatment Follow-up Period (N=210)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weeks 1 to 14: Dapagliflozin 5 mg (N=81) | Weeks 14 to 26: Dapagliflozin 5 mg (N=55) | Weeks 14 to 26: Dapagliflozin 10 mg (N=21) | Weeks 26 to 56: Dapagliflozin 5 mg (N=55) | Weeks 26 to 56: Dapagliflozin 10 mg (N=21) | Weeks 32 or 40 to 56: Dapagliflozin 10 mg + Metformin Withdrawal (N=7) | Weeks 1 to 14: Saxagliptin 2.5 mg (N=88) | Weeks 14 to 26: Saxagliptin 2.5 mg (N=61) | Weeks 14 to 26: Saxagliptin 5 mg (N=26) | Weeks 26 to 56: Saxagliptin 2.5 mg (N=61) | Weeks 26 to 56: Saxagliptin 5 mg (N=26) | Weeks 32 or 40 to 56: Saxagliptin 5 mg + Metformin Withdrawal (N=13) | Weeks 1 to 14: Placebo (N=76) | Weeks 14 to 26: Placebo (N=70) | Weeks 26 to 32 or 40: Placebo (N=70) | Weeks 32 or 40 to 56: Placebo (N=53) | Weeks 32 or 40 to 56: Placebo to Dapagliflozin 10 mg + Metformin Withdrawal (N=3) | Weeks 32 or 40 to 56: Placebo to Saxagliptin 5 mg + Metformin Withdrawal (N=3) | Week 56 to 104: Non-treatment Follow-up Period (N=210)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Albumin urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial test (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose normal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood parathyroid hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Primary hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-telopeptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mean cell haemoglobin concentration decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mean cell haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 5 (5) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premenstrual pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sphenoid sinus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balanitis candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal balanitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericoronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wolff-parkinson-white syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Closed globe injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to legal dispute, the source documents could not be accessed for 11 participants at 1 site. All data from this site were excluded as documented in the statistical analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03199053/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03199053/SAP_003.pdf